CLINICAL TRIAL: NCT04161014
Title: The Nintedanib in Progressive Pneumoconiosis Study (NiPPS): a Collaborative NSW Treatment Trial
Acronym: NiPPs
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Holdsworth House Medical Practice (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Deborah Yates, Associate Professor Deborah Yates, Holdsworth House Medical Practice
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NiPPs
Record Dates: First submitted 2019-11-07; First posted 2019-11-13 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Pneumoconiosis Coal; Asbestosis; Silicosis
MeSH Terms: conditions — Anthracosis; Asbestosis; Silicosis | interventions — nintedanib

STUDY DESIGN:
Intervention Model Description: Prospective clinical pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Other): Nintedanib 150mg twice daily for 3 years
  Interventions: Drug: Nintedanib 150 MG [Ofev]

INTERVENTIONS:
Drug: Nintedanib 150 MG [Ofev] — Nintedanib 150mg twice daily for 3 years

SUMMARY:
Prospective clinical pilot study for subjects diagnosed with Occupational Progressive Pneumoconiosis.

Subjects will be treated with Nintedanib 150mg twice daily for 3 years.

DETAILED DESCRIPTION:
100 Patients with asbestosis, silicosis, coal workers pneumoconiosis and diffuse dust fibrosis will be included. Patients will have an FVC ≥45% predicted (no upper threshold), and a diffusion capacity of the lung for carbon monoxide (TLCO) above 30% predicted. Patients will be randomised to receive Nintedanib 150 mg twice daily, with the dose of the study drug reduced to 100 mg twice daily or interrupted temporarily in the case of adverse events (AEs).The primary end point will be the annual decline in FVC, measured in millilitres per year, calculated from serial measurements over 36 months.

Lung function testing will be performed at baseline; 2, 4, 6, 12, 18, 24, 30, 36, 44 and 52 weeks, and every 4 months thereafter until study cessation or withdrawal at a maximum of 36 months.

In patients who show clinical benefit as per the end points specified access to Nintedanib treatment will be continued.

ELIGIBILITY:
Inclusion Criteria:

* Pneumoconiosis diagnosis confirmed at the Occupational MDT (Occ-MDT)
* diffuse fibrosing lung disease of extent >10% on HRCT with protocol criteria for progression
* Asbestosis, silicosis, coal worker's pneumoconiosis and diffuse dust fibrosis
* FVC ≥45% predicted and TLCO above 30% predicted

Exclusion Criteria:

* idiopathic pulmonary fibrosis (IPF) and non-occupational progressive pulmonary fibrosis
* ILD due to connective tissues disorders, hypersensitivity pneumonitis, non-occupational interstitial pneumonia, non-occupational sarcoidosis
* contraindications to Nintedanib (forthcoming surgery, use of anticoagulants, high CVD risk, liver function abnormalities)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-09 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
annual decline in FVC | 36 months
  measured in millilitres per year, calculated from serial measurements

SECONDARY OUTCOMES:
K-BILD score | week 52
  Absolute change from baseline in King's Brief Interstitial Lung Disease Questionnaire (K-BILD) total score. The KBILD domain and total score ranges are 0-100; 100 represents best health status
Time to acute exacerbation | 36 months
  an acute, clinically significant respiratory deterioration characterized by evidence of new, widespread alveolar abnormality, including unexplained worsening or development of dyspnea,new diffuse pulmonary infiltrates visualized on chest radiography, HRCT, or both, or the development of parenchymal abnormalities with no pneumothorax or pleural effusion (new ground-glass opacities) since the preceding visit; and exclusion of any known causes of acute worsening, including infection, left heart failure, pulmonary embolism, and any identifiable cause of acute lung injury, in accordance with routine clinical practice and microbiologic studies.
Time to referral for Lung transplantation | 36 months
  Respiratory deterioration which necessitates a referral for lung transplant
Time to death | 12, 24 and 36 months
  Respiratory deterioration leading to death

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Yates, A/Prof, Principal Investigator — Holdsworth House Medical Practice
Locations (1):
- Holdsworth House Medical Practice, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No